CLINICAL TRIAL: NCT01790022
Title: Efficacy and Safety of MEthylprednisolone Administered Intravenously for the Treatment of Patients With Active AnkyLosing spondyLitis (METALL) - a 12-week, Prospective, Open-label, Pilot Study
Brief Title: Efficacy and Safety of MEthylprednisolone Administered Intravenously for the Treatment of Patients With Active AnkyLosing spondyLitis (METALL)
Acronym: METALL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Saratov State Medical University (Other)
Collaborators: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Denis Poddubnyy, MD, Saratov State Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: METALL 2012
Record Dates: First submitted 2013-02-09; First posted 2013-02-12 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2013-02

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Methylprednisolone; Methylprednisolone Hemisuccinate

ARMS (1):
- Methylprednisolone 500 mg (Experimental): Methylprednisolone 500 mg administered intravenously at baseline
  Interventions: Drug: Methylprednisolone

INTERVENTIONS:
Drug: Methylprednisolone
  Other Names: Metypred, Medrol, Solu-Medrol

SUMMARY:
In this study, efficacy of methylprednisolone in reduction of signs and symptoms (back pain, stiffness, joint pain and swelling) of active ankylosing spondylitis (AS) will be investigated. It is expected, that a single dose of methylprednisolone 500 mg given intravenously at baseline will lead to a rapid reduction of symptoms of active AS, which can be seen already 2 weeks after drug administration.

ELIGIBILITY:
Inclusion Criteria:

* Age of ≥18 years.
* Definite diagnosis of AS according to the modified New York criteria.
* History of an inadequate response to ≥2 nonsteroidal antiinflammatory drugs (NSAIDs) taken for at least 2 weeks each or NSAIDs intolerance.
* Active disease as defined by the Bath Ankylosing Spondylitis DIsease Activity Index (BASDAI) value of ≥4 at screening despite concomitant treatment with an NSAID or without NSAIDs in case of intolerance.

Exclusion Criteria:

* The female subject is pregnant or lactating.
* Patients with other chronic inflammatory articular disease or systemic autoimmune disease.
* History of inadequate response to previous anti-tumour necrosis factor (TNF) α therapy.
* Treatment with any other investigational drug within 4 weeks of 5 half-life of the drug (whichever is longer) prior to baseline.
* Treatments with disease modifying anti-rheumatic drugs (DMARDs) other than methotrexate within 4 weeks prior to screening (8 weeks for leflunomide or 4 weeks with a standard cholestyramine wash-out).
* Treatment with intravenous, intramuscular or intraarticular/periarticular steroids within 4 weeks prior to screening.
* History of oesophageal, gastric, duodenal or intestinal ulceration, clinically relevant gastrointestinal bleeding.
* History of or current signs of coronary heart disease, myocardial infarction, stroke or transient ischemic attack, peripheral arterial thrombotic events.
* Congestive heart failure (NYHA III-IV)
* Uncontrolled arterial hypertension.
* History of diabetes mellitus.
* History of glaucoma.
* Major surgery within 12 weeks prior to screening.
* Evidence of any other severe uncontrolled gastrointestinal, hepatic, renal, pulmonary, cardiovascular, nervous or endocrine disorders.
* Any active current viral, bacterial or fungal infection, a history of recurrent clinically significant infection, infections requiring treatment with antibiotics within 4 weeks prior to baseline.
* History of chronic infection with hepatitis B or C, history of HIV infection.
* Primary or secondary immunodeficiency.
* Any other conditions making the patient unsuitable in the opinion of the investigator for the participation in the current study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-07; Primary Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
The Assessment of Spondyloarthritis International Society 40 (ASAS40) response | Week 2
  The Assessment of Spondyloarthritis International Society 40 (ASAS40) response is defined as an improvement of ≥40% and ≥2 points in at least 3 out of four following domains (and no worsening in remaining domain):
  * Patient global
  * Pain
  * Function (as measured by the Bath Ankylosing Spondylitis Functional Index - BASFI)
  * Inflammation (mean of the Bath Ankylosing Spondylitis Disease Activity Index - BASDAI question 5 and 6)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Rheumatology, Saratov Region Hospital, Saratov, Russia